CLINICAL TRIAL: NCT01027065
Title: A Phase Randomized Open Labelled Controlled Dose Escalation Study of Repeated Administration of "CYT107" (Glyco-r-hIL-7) Added on Antiviral Treatment and Vaccination in HBeAg-negative Chronic Hepatitis B-infected Patients
Brief Title: Dose Escalation of Interleukin-1 (IL-7) Added on Antiviral Treatment and Vaccination in HBeAg-negative Chronic Hepatitis B Virus (HBV) Infected Patients
Acronym: CONVERT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cytheris SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLI-107-10; 2009-010709-35 (Other: EUDRACT Number)
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Hepatitis B
Keywords: interleukin-7; immune-based therapies; hepatitis B; HBe negative; HBV vaccination; entecavir; tenofovir; chronic hepatitis; immune specific responses to HBV; phase 1/2a; viral disease; liver disease
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B; Hepatitis, Chronic; Virus Diseases; Liver Diseases | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tritherapy: CYT107+ vaccine+ antiviral (Experimental)
  Interventions: Drug: CYT107+GenHevac+entecavir or tenofovir
- Bitherapy: CYT107 + antiviral (Experimental)
  Interventions: Drug: CYT107+ entecavir or tenofovir

INTERVENTIONS:
Drug: CYT107+GenHevac+entecavir or tenofovir — 4 patients per arm for each dose level. 3 patients receiving experimental treatment (CYT107 and vaccine) in addition to current antiviral treatment and 1 control patient only the current antiviral treatment
  Arms: Tritherapy: CYT107+ vaccine+ antiviral
Drug: CYT107+ entecavir or tenofovir — 4 patients per arm for each dose level. 3 patients receiving experimental treatment (CYT107) in addition to current antiviral treatment and 1 control patient only the current antiviral treatment
  Arms: Bitherapy: CYT107 + antiviral

SUMMARY:
This study is designed to evaluate the safety of biological active dose of a new experimental drug, IL-7, in combination with anti viral therapy and vaccine in patients with Hepatitis B chronic infection.

DETAILED DESCRIPTION:
This is a Phase I/IIa inter-patient dose-escalation study assessing weekly doses of Interleukin-7 (CYT107) in HBeAg-negative chronic hepatitis B infected adult patients. The dose escalation is aimed at establishing the safety of a biologically active doses of CYT107 added to the current antiviral therapy with entecavir or tenofovir and vaccination or not. At each dose level, study patients will receive one subcutaneous administration of CYT107 per week for a total of 4.

Groups of 8 patients will be entered at each dose level of CYT107. Three dose levels are planned.

At each dose level, patients are randomized between 2 arms of treatment: tritherapy (CYT107, vaccine and antiviral treatment) or bitherapy (CYT107 and vaccine). Each treatment group is composed of 4 patients, 3 receiving experimental treatments, 1 just the current antiviral treatment (control patient).

According to the treatment arm, eligible patients initially receive a vaccine if in treatment group of tritherapy, thereafter, CYT107 is added for a cycle of four weekly injections (if not a control patient) at a defined dose level. If in treatment group of tritherapy, patients will receive 2 additional doses of vaccine.

The treatment phase for the tritherapy group is from first vaccine D0 to last vaccine W12 and includes CYT107 administration from W4 to W7.

The treatment phase for the bitehrapy group is from W4 to W7 corresponding to CYT104 injections.

The patients are then followed on a regular basis until reaching 52 weeks after the D0.

Participants will have 1 overnight hospitalization and 12 clinic visit on a period of 55 weeks.

During the visits the following may be done:

* medical history, physical examination, blood tests
* electrocardiograms (ECG)
* chest X-Ray
* liver/spleen imaging
* urine tests

ELIGIBILITY:
Inclusion Criteria:

* Chronic HBV-infected patients
* HBeAg-negative patients
* Age > 18 years
* Patients with active chronic hepatitis at the start of the antiviral treatment
* Patient with a HBV DNA undetectable (<70 copies/ml) stable for at least 3 months under entecavir or tenofovir treatment.
* Ongoing treatment by entecavir or tenofovir at screening Note: previous treatment with pegylated IFN monotherapy, before the start of entecavir or tenofovir, is acceptable

Exclusion Criteria:

* Infection by HCV
* Infection by HIV-1 and /or HIV-2
* Apart from HBV infection, presence of active infection requiring a specific treatment or a hospitalization
* Previous treatment by lamivudine and/or nucleosides analogues
* Inactive carrier
* Cirrhosis
* Other liver disease (notably from alcoholic, metabolic or immunological origin)
* History of clinical autoimmune disease or active auto-immune disease
* Type I diabetes mellitus
* Severe asthma, presently on chronic medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-12; Primary Completion 2012-11 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
To determine the short and long-term safety and biological activity of CYT107 in patients with a HBeAg-negative chronic hepatitis B who have, at screening a HBV DNA undetectable stable for at least 3 months with antiviral treatment. | Week 12

SECONDARY OUTCOMES:
To characterize the pharmacokinetics and pharmacodynamics of CYT107 in humans chronically infected with HBV. | Week 12
To assess the effects of the tri-therapy (CYT107 + HBV vaccine + antiviral treatment) versus bi-therapy (CYT107 + antiviral treatment) versus control (antiviral treatment) on the markers of the HBV infection (antiviral activity)at W16 weeks and W52 | Week 12 and Week 52
To quantify the effects of the tri-therapy (CYT107 + HBV vaccine + antiviral treatment) versus bi-therapy (CYT107 + antiviral treatment) versus control (antiviral treatment) on the immune system at W16 weeks | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Hezode, Study Chair — Hopital Henri Mondor-Créteil-France; Pietro Andreone, Principal Investigator — S. Orsola Malpighi- Bologna-Italy
Locations (8):
- France (7):
  - Hopital Henri Mendor-Service d'HepatoGastroEnterologie, Créteil
  - Hopital Michallon, Grenoble
  - Hopital de l'Hotel Dieu, Lyon
  - Hopital Saint Joseph, Marseille
  - CHU l'Archet, Nice
  - Hopital Tenon, Paris
  - Hopital Civil, Strasbourg
- Azienda Ospedaliero-Universitaria, Policlinico Sant'Orsola Malpighi, Bologna, Italy